CLINICAL TRIAL: NCT05646472
Title: Approccio Multidimensionale Supportato Dalle ICT Per lo Screening Della fragilità Nei Soggetti di età ≥ 65 Anni Che Vivono in comunità - SUNFRAIL+
Brief Title: ICT-supported Multidimensional Approach for Frailty Screening in Community-dwelling Individuals Aged ≥ 65 Years
Acronym: SUNFRAIL+
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Maddalena Illario, Prof, Federico II University
Other Study IDs: 284/22
Record Dates: First submitted 2022-12-01; First posted 2022-12-12 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Frail Elderly Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ≥ 65 Community-dwelling older adults
  Interventions: Diagnostic Test: Frailty multidimensional assessment

INTERVENTIONS:
Diagnostic Test: Frailty multidimensional assessment — Each Centre will administer SUNFRAIL frailty assessment tool to the enrolled older adults and, according to the specific "alerts" triggered by the answers provided, older adults will be subjected (at the same time or subsequently) to one or more validated in-depth tests (already included in the SUNFRAIL+ platform) in order to perform further diagnostic or dimensional evaluations.
  During the observation phase, subjects will be given different health promotion activities, depending on the assessment.
  During the follow-up phase, 6 months after enrolment, SUNFRAIL tool and in-depth tests will be administered again. In addition, during the follow up, the extent to which exposure to interventions has influenced the quality of life of older adults will be measured and the number of users enrolled by territorial services, based on user care needs. In addition, the level of satisfaction and usability of the SUNFRAIL+ solution by health and social care professionals will be measured.

SUMMARY:
SUNFRAIL+ is a prospective observational cohort study aimed to carry out a multidimensional assessment of community-dwelling older adults, through an IT platform, which allows to connect the items of the SUNFRAIL frailty assessment tool with a cascading multidimensional in-depth assessment of the bio-psycho-social domains of frailty. It is a multicentric study. Seven centres will administer SUNFRAIL questionnaire to 100 older adults each and, according to the specific "alerts" triggered by the answers provided, older adults will be subjected to one or more validated in-depth tests in order to perform further diagnostic or dimensional evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years;
* Living at home;
* accessing participating centres for social and healthcare services other than those covered by this study;
* ability to sign the informed consent

Exclusion Criteria:

* Age <65 years;
* Residents in care facilities (hospital, nursing home);
* have overt frailty or disability; are already enrolled in home care; are unable to understand the study aims and sign the informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: primary care clinic, community sample
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Improved quality of life | Month 14
  Impact of early, integrated and simultaneous "taking care" by health system on the quality of life of community-dwelling older adults
Appropriateness of care | Month 14
  Level of appropriateness of care by the healthcare system
Level of satisfaction of the health professionals | Month 14
  Impact of the IT solution on the organization of services and the workload of professionals

CONTACTS AND LOCATIONS:
Locations (8):
- Italy (8):
  - Azienda Socio Sanitaria Territoriale della Valle Olona, Busto Arsizio
  - Azienda Sanitaria Locale Cuneo 1, Cuneo
  - Azienda Sociosanitaria Ligure n. 4, Genova
  - Azienda Unità Sanitaria Locale Nord-Ovest, Lucca
  - Azeidna Ospedaliera Universitaria Federico II, Napoli
  - Cooperativa Sociale "Res Omnia", Reggio Calabria
  - Dipartimento di Biomedicina e Prevenzione dell'Università degli Studi di Roma Tor Vergata, Roma
  - Azienda Provinciale Socio-Sanitaria Trento, Trento

IPD SHARING:
Plan to Share IPD: Yes
Study protocol will be published on an open access scientific journal
Supporting Information: Study Protocol

REFERENCES:
- [Derived] De Luca V, Femminella GD, Leonardini L, Patumi L, Palummeri E, Roba I, Aronni W, Toccoli S, Sforzin S, Denisi F, Basso AM, Ruatta M, Obbia P, Rizzo A, Borgioli M, Eccher C, Farina R, Conforti D, Mercurio L, Salvatore E, Gentile M, Bocchino M, Sanduzzi Zamparelli A, Viceconte G, Gentile I, Ruosi C, Ferrara N, Fabbrocini G, Colao A, Triassi M, Iaccarino G, Liotta G, Illario M. Digital Health Service for Identification of Frailty Risk Factors in Community-Dwelling Older Adults: The SUNFRAIL+ Study Protocol. Int J Environ Res Public Health. 2023 Feb 21;20(5):3861. doi: 10.3390/ijerph20053861. PMID 36900872